CLINICAL TRIAL: NCT05198921
Title: The Effectiveness of Repetitive Transcranial Magnetic Stimulation for the Treatment of Spastic Diplegia Cerebral Palsy Based on the Gross Motor Function in School-aged Children: a Randomized Controlled Trial
Brief Title: The Effectiveness of Repetitive Transcranial Magnetic Stimulation for Spastic Diplegia Cerebral Palsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Clàudia Arumí, Principal Investigator, Universitat de Lleida
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ULleida1
Record Dates: First submitted 2021-12-27; First posted 2022-01-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Palsy, Spastic
MeSH Terms: conditions — Cerebral Palsy | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: randomized crossover double-blind trial. It is a pre-post study with follow-up at 1 month
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rTMS + neurorehabilitation (Experimental)
  Interventions: Device: repetitive Transcranial Magnetic Stimulation; Device: sham repetitive Transcranial Magnetic Stimulation
- sham rTMS + neurorehabilitation (Sham Comparator)
  Interventions: Device: repetitive Transcranial Magnetic Stimulation; Device: sham repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation — To apply the rTMS will be used the device Neuro-MS/D Variant-3 therapeutic advanced (Neurosoft, Russia) with double cone shape coil. The coil will be placed at Cz according to 10-20 system.
  The rTMS protocol will be:
  Train frequency - 10 Hz Train duration - 10 sec Inter train interval - 50 seconds Number of train - 25
  ------------------------------------- Total pulses - 2500 Total session duration - 1500 seconds
Device: sham repetitive Transcranial Magnetic Stimulation — Neuro-MS/D magnetic stimulator (Neurosoft, Russia) with Neuro-MS.NET software will be used. The synchronous sound will be performed using monitor speaker connected to magnetic stimulator via trigger unit and located near discharging coil. The 10-Hz electrical stimulation will be given trough electrodes fixed on the head along the front edge of the coil to mimic the sensation

SUMMARY:
Cerebral palsy describes a group of permanent disorders of the development of movement and posture, causing activity limitation that are attributed to non-progressive disturbances that occurred in the developing fetal or infant brain.

Nowadays, CP is not fully curable, and physiotherapy should be used in conjunction with other interventions such as oral drugs, botulinum toxin type A, continuous pump-administered intrathecal baclofen, orthopaedic surgery and selective dorsal rhizotomy. However, several systematic reviews conclude that there is low evidence that these invasive therapies are more effective than placebo.

Repetitive transcranial magnetic stimulation (rTMS) is a type of neuromodulatory technique through magnetic impulses. The effect of rTMS depends on the frequency of the emitted electromagnetic field; low frequencies (≤1 Hz) lead to an inhibition of neuronal electrical activity at the stimulation site, while high frequencies (≥3 Hz) cause neuronal depolarization.

The objective of the project is to evaluate the effectiveness of a repetitive Transcranial Magnetic Stimulation (rTMS) protocol, as an adjunct treatment to neurorehabilitation to improve gross motor function and quality of life in school-age children with spastic diplegia-type infantile cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy describes a group of permanent disorders of the development of movement and posture, causing activity limitation that are attributed to non-progressive disturbances that occurred in the developing fetal or infant brain.

The reported worldwide prevalence rates of CP are approximately between 2 and 3 per 1000 live births. In Spain, it is estimated that between 2 and 2.5 per thousand born has cerebral palsy, that is, 1 per in 500 live births. In other words, in Spain there are 120,000 people with cerebral palsy.

The Spastic Diplegia form is the most common form with around 65-70 % of the CP children. It is characterized by gross motor difficulties, marked in the lower limb and partially affection noticeable in the upper limb.

Spasticity is defined as "disordered sensori-motor control, resulting from an upper motoneuron lesion, presenting as intermittent or sustained involuntary activation of muscles". Spasticity is a velocity-dependent motor disorder, characterized by an increased stretch reflex, resulting in immoderate muscle activation that causes a muscle hypertonia. The pathophysiology of spasticity is characterized, in general, by a deregulation of the motor pathways (mainly the corticospinal, reticulospinal, and the vestibulospinal tracts) running from the cerebral cortex, and brain stem to the spinal cord. In children who suffer from an early brain abnormality, spasticity is affected by the reorganization of supraspinal input and impaired motor maturation, causing a loss in descending inhibitory inputs and an increase of the excitability of gamma and alpha neurons.

NICE clinical guidance recommends the use of physiotherapy, as it provides an approach centred on how the current functional problems impact on the participation at home, school life and community. Nowadays, CP is not fully curable, and physiotherapy should be used in conjunction with other interventions such as oral drugs, botulinum toxin type A, continuous pump-administered intrathecal baclofen, orthopaedic surgery and selective dorsal rhizotomy. However, a recent Cochrane Systematic Review (CSR) concludes that there is low evidence that BoNT-A is more effective than placebo or a non-placebo control in children with CP. Another recent CSR determines that there is short-term evidence of the Intrathecal Baclofen therapy. Furthermore, there is not a CSR for orthopaedic surgery and selective dorsal rhizotomy.

Non-invasive brain stimulation Repetitive Transcranial Magnetic Stimulation (rTMS) is a type of neuromodulator technique in which trains are emitted from multiple magnetic pulses. The effect of rTMS depends on the emitted electromagnetic field frequency; low frequencies (≤1 Hz) lead to an inhibition of neural electrical activity at the stimulation site, while high frequencies (≥3 Hz) cause neuronal depolarization. It has been reported that rTMS stimulation of prefrontal and motor cortical areas gives rise to trans synaptic activation of subcortical circuits which are responsible for motor activity and reduction of muscle spasticity. That is, an increase in the activity in the motor cortex, increases the inhibitory input to the corticospinal tract and reduces the hyperactivity of the gamma and alpha neurons.

In terms of scientific evidence, some researchers have already studied the effect of rTMS over standard therapy in decreasing muscle tone in CP patients, such as Gupta et al. who demonstrated better results on the group who carried out the treatment compared to the control group. Lal Rajak et al. studied how the number of therapy sessions of rTMS would improve the motor development by reducing muscle spasticity in children with CP, and concludes that the group which carried out more sessions, showed better improvements. Gupta and Lal Rajak also studied the efficacy of different pulses by a constant frequency. They found that in diplegic patient's, the gross motor function improved by 3.04%, 4.62% and 5.95% in groups of 1500 pulses, 2000 pulses and 2500 pulses, respectively.

However, all the randomized controlled trials (RCTs) conducted as of yet, showed limitations on the methodological quality. They all presented a very small sample size, which makes difficult to conclude that the therapy is effective. Moreover, neither did an evaluation in the middle of the treatment, only at the beginning and at the end, so it is not known if the therapy begins to produce effect sooner, and none of them conducted long-term monitoring results. Additionally, they only used one evaluation measure, the Modified Ashworth scale. Besides, none of the RCTs took into account the family or carers, which have a main role on making decisions and care planning.

ELIGIBILITY:
Inclusion Criteria:

* Primary school children with diagnose of Spastic Diplegia CP
* > 1 on Mas in hip flexors, adductors and tibialis anterior of both lower extremities.
* Parents/legal guardians signed the Informed consent

Exclusion Criteria:

* Severe mental retardation
* Present epilepsy
* Present any remedial surgery/medication
* Less than 1 year post orthopaedic surgery
* Less than 6 months post botulinum toxin type A injection
* Present metallic implants
* Present any comorbidity unfit for the study
* Congenital disorders such as Down's syndrome, fragile-x syndrome or congenital anomalies

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in Gross Motor Function by the Gross Motor Function-66 | baseline, one month, two months, three months and six months.
  The GMFM is a standardized assessment instrument designed to measure change over time in gross motor function in cerebral palsy children. The GMFS-66 is an 66-item measure with five dimensions: lying and rolling, crawling/kneeling, standing and walking/running/jumping. Each GMFM item is graded on a 4-point scale. The magnitude of change that is considered clinically important for an individual child will vary and depend on the judgments made by the child, family, and therapist. It takes between 20-25 minutes to be completed. GMFM presents good longitudinal construct validity, the test - retest is high with a 0.99 ICC and researchers indicate that GMFM adequately measure change over time in gross motor function for children with CP.

SECONDARY OUTCOMES:
Change in Functional Strength by the Functional Strength Measure | baseline, one month, two months, three months and six months.
  The functional strength measurement (FSM) measures functional strength in both, upper and lower extremities. It consists of eight items matching activities of children in aged group from 4 to 10 years with typically developing (TD). The FSM has been adapted for children with CP (FSM-CP). The test-retest reliability of FSM-CP, has shown to be high and the comparison of the scores on the FSM-CP with the HHD showed mostly moderate correlations. In the present study, only the items related to lower extremities will be evaluated. Participants will have the opportunity to practice every test item maximum five trials before being tested. Each item will be examined three times and the highest score will be the useful for the analysis. To be able to say that a child improved after a treatment, needs to improve his/her score from the last examination.
Change in Quality of Life by the Cerebral Palsy Quality of Life-Child | baseline, one month, two months, three months and six months.
  The CP QOL-Child is questionnaire designed to assess the QOL in children aged between 4-12 years. It is composed by two parts. The first one a caregiver/parent report for children aged 4 to 12 years and the second one is a self-report of children aged from 9 to 12 years. The parent-proxy version comprises 65 items, and the child self-report version comprises 53 items. The CP QOL-Child measures the seven areas of child's life such as; social wellbeing and acceptance, participation and physical health, feelings about functioning, emotional wellbeing and self-esteem, pain and impact of disability, access to services, and family health. For each question there's a number 1 (very unhappy) to 9 (very happy) (46). The scoring involves two steps. At the first step the items are transformed to a scale with a possible range of 0-100 and the second step it is done by the algebraic mean of item values for each domain. The scoring process is explained on the CP QOL-Child manual 2nd version.
Change in Spasticity by the Modified-Modified Ashworth Scale. | baseline, one month, two months, three months and six months.
  The scale most commonly used to evaluate spasticity is the Ashworth scale (AS) and the Modified Ashworth Scale (MAS). The ICC scores of interrater reliability ranged from 0.54 to 0.80 and the intrarater reliability from 0.31 to 0.82. MAS is the primary outcome measure but at the time of data analysis the grades are modified (m-MAS), Modified-Modified Ashworth Scale. Therefore, the Rehabilitation Measures Database, suggests that a one-point change on the MAS reflects a clinically significant improvement. The score is based on the resistance felt during that one second of passive movement and it should be done 1-3 times at most. The target muscles will be hip flexors, adductors and tibialis anterior in both lower extremities. Physiotherapists will be experienced in applying MAS.
Change in Impact on family by the Revised Impact on Family questionnaire | baseline, one month, two months, three months and six months.
  The RIOF scale was designed specifically to measure the impact of paediatric chronic illness on the family. It consists of 15 items with good psychometric properties. Each item represents a statement about having a chronically ill or disabled child. Parents/legal guardians are asked to rate on a four-level scale (strongly disagree or strongly agree) to which degree each of the items applies to the current situation of the family. The instrument is also reliable and valid to be implemented with chronic hospitalized children.
Cortex excitability | Enrollment, 1st month, 2nd month, 3rd month and 4th month
  Motor cortex excitability will be measured using a magnetic stimulator with a figure-eight coil. Responses to stimuli applied to motor cortices will be recorded in the adductor muscles and the hip flexors in both lower limbs.

CONTACTS AND LOCATIONS:
Locations (1):
- Claudia Arumi, Lleida, Lleida, Spain

IPD SHARING:
Plan to Share IPD: No